CLINICAL TRIAL: NCT05438901
Title: Investigation of Oxidant-antioxidant Status in Patients Treated With Hirudotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, İsmail Sarıkan, Asst. Prof. Dr.(MD, PhD), Alanya Alaaddin Keykubat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 123ism456kny
Record Dates: First submitted 2022-03-26; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Leeches
Keywords: Hirudotherapy; leech therapy; total antioxidative status; total oxidative status
MeSH Terms: interventions — Leeching

STUDY DESIGN:
Intervention Model Description: A single-group study was conducted before (1st arm) and after (2nd arm) administration of HT.
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- before and after application (Experimental): Before the hirudotherapy application, it was planned to study the oxidant and antioxidant parameters in the venous blood of the patient. In addition, it was planned to study the oxidant and antioxidant parameters in the patient's venous blood after 2 sessions of Hirudotherapy, 1 month apart.
  Interventions: Biological: leech therapy

INTERVENTIONS:
Biological: leech therapy — effects of medicinal leeches

SUMMARY:
Hirudotherapy (HT); It is a traditional treatment method applied using medicinal leeches such as Hirudo Medicinalis and Hirudo Verbana.

Purpose of the study titled "Investigation of oxidant-antioxidant status in patients treated with hirudotherapy": To investigate the effect of HT on oxidative stress in healthy individuals.

DETAILED DESCRIPTION:
Ethics committee decision dated 14.08.2020 and numbered 22-40 was taken from Alanya Alkü Medical Faculty Clinical Research Ethics Committee. Participants will be accepted into the study after signing and approving the informed consent form (ICF). All procedures performed in studies involving human participantswere in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards.

This study will be carried out at Alanya Training and Research Hospital Traditional and Complementary Medicine (Getat) Application Center between 29 March-29 September 2021 with fifty (50) volunteers. All participants will receive hirudotherapy twice, 1 month apart. Venous blood samples will be taken before the first application (pre-HT) and after the second application (post-HT), total antioxidant capacity (TAS) and total oxidant capacity (TOS) in the serum portion of the blood samples taken, as well as oxidative stress index (OSI=TOS/TAS), ischemia modified albumin (IMA), paraoxonase 1 (PON1), disulfide, natural thiol, total thiol, arylesterase (ARES) will be measured. The above biochemical parameters will be investigated in serum using fully automatic colorimetric methods.

Statistical analyzes of the data were performed using the SPSS 15.0 program (SPSS Inc. and Lead Tech. Inc. Chicago. USA). The significance of the difference between the two groups was evaluated with the Independent samples t test, which is a parametric method. Data are presented as mean ±SD. In the statistical evaluation, p<0.05 was considered significant.

Limitations of this study: 1) No control group, 2) No dietary restriction between sessions (For example, not limiting the intake of foods known to have antioxidant effects, etc.). The strength of this study is that it is supported by the scientific research projects coordinatorship of the university, which is an impartial financial resource.

Financial support: This study was financially supported by Alanya Alaaddin Keykubat University (Alkü) Scientific Research Projects Coordinatorship with project number 2021-04-02-MAP10.

ELIGIBILITY:
Exclusion criteria for the study:

1. Bleeding diathesis (such as hemophilia)
2. Pregnancy and breastfeeding status
3. History of allergy to leech
4. Age under 18

Inclusion criteria for the study:

1) Not have an active bleeding problem

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 30 women and 20 men
Enrollment: 12317546 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Examination of the change in biochemical parameters from the beginning, TAS sample | From baseline to 0-3 months and 3-6 months
  Biochemical parameters will be measured by fully automatic colorimetric method in Alaaddin Keykubat University Faculty of Medicine Biochemistry Laboratory. TAS(Total anti-oxidant status), Unit: mmol Trolox Eq/L.Function: It is a method that measures the total antioxidant capacity of the body.
Examination of the change in biochemical parameters from the beginning, TOS sample | From baseline to 0-3 months and 3-6 months
  Biochemical parameters will be measured by fully automatic colorimetric method in Alaaddin Keykubat University Faculty of Medicine Biochemistry Laboratory. TOS(Total oxidant status), Unit:μmol H2O2 Eq/L, Function: It is a colorimetric method that measures the total oxidant capacity of the body that occurs in metabolic processes.

CONTACTS AND LOCATIONS:
Overall Officials: ismail sarikan, Asst.Prof., Principal Investigator — Alaaddin Keykubat University
Locations (1):
- Alaaddin Keykubat University, Alanya, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Tagil SM, Celik HT, Ciftci S, Kazanci FH, Arslan M, Erdamar N, Kesik Y, Erdamar H, Dane S. Wet-cupping removes oxidants and decreases oxidative stress. Complement Ther Med. 2014 Dec;22(6):1032-6. doi: 10.1016/j.ctim.2014.10.008. Epub 2014 Oct 13. PMID 25453524
- [Background] Godekmerdan A, Arusan S, Bayar B, Saglam N. [Medicinal leeches and hirudotherapy]. Turkiye Parazitol Derg. 2011;35(4):234-9. doi: 10.5152/tpd.2011.60. Turkish. PMID 22198928
- [Result] Erel O, Neselioglu S. A novel and automated assay for thiol/disulphide homeostasis. Clin Biochem. 2014 Dec;47(18):326-32. doi: 10.1016/j.clinbiochem.2014.09.026. Epub 2014 Oct 7. PMID 25304913
- [Result] Gultekin F, Naziroglu M, Savas HB, Cig B. Calorie restriction protects against apoptosis, mitochondrial oxidative stress and increased calcium signaling through inhibition of TRPV1 channel in the hippocampus and dorsal root ganglion of rats. Metab Brain Dis. 2018 Oct;33(5):1761-1774. doi: 10.1007/s11011-018-0289-0. Epub 2018 Jul 16. PMID 30014177
- [Result] Sies H, Berndt C, Jones DP. Oxidative Stress. Annu Rev Biochem. 2017 Jun 20;86:715-748. doi: 10.1146/annurev-biochem-061516-045037. Epub 2017 Apr 24. PMID 28441057
- [Result] Valko M, Leibfritz D, Moncol J, Cronin MT, Mazur M, Telser J. Free radicals and antioxidants in normal physiological functions and human disease. Int J Biochem Cell Biol. 2007;39(1):44-84. doi: 10.1016/j.biocel.2006.07.001. Epub 2006 Aug 4. PMID 16978905
- See also: Related Info — http://www.who.int/health-topics/traditional-complementary-and-integrative-medicine
- See also: Related Info — http://shgmgetatdb.saglik.gov.tr